CLINICAL TRIAL: NCT00986609
Title: Pilot Study of a MUCI Peptide and Poly-ICLC Vaccine for Triple-Negative Breast Cancer
Brief Title: MUC1 Vaccine for Triple-negative Breast Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Joseph Baar, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Joseph Baar, MD, PhD, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CASE16107; NCI-2009-01318 (Other: NCI/CTRP)
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Breast Cancer; Inflammatory Breast Cancer; Stage I Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Triple-negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — poly ICLC; Enzyme-Linked Immunosorbent Assay; Flow Cytometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive MUC-1 peptide vaccine subcutaneously and poly-ICLC vaccine intramuscularly in weeks 0, 4, 8, 12, 52, and 56, in the absence of disease progression or unacceptable toxicity. Patients may receive additional vaccines in weeks 34 and 38 if anti-MUC1 immunity falls below the two-fold enhancement from baseline
  Interventions: Biological: MUC-1 peptide vaccine; Biological: poly ICLC; Biological: MUC1 peptide-poly-ICLC adjuvant vaccine; Other: laboratory biomarker analysis; Other: enzyme-linked immunosorbent assay; Other: flow cytometry

INTERVENTIONS:
Biological: MUC-1 peptide vaccine — Given subcutaneously
Biological: poly ICLC — Given intramuscularly
  Other Names: Hiltonol; poly I:poly C with poly-1-lysine stabilizer; Polyinosinic-Polycytidylic Acid Stabilized with Polylysine and Carboxymethylcellulose; Polyriboinosinic-Polyribocytidylic Acid-Polylysine Carboxymethylcellulose; stabilized polyriboinosinic/polyribocytidylic acid
Biological: MUC1 peptide-poly-ICLC adjuvant vaccine — Receive adjuvant vaccination
Other: laboratory biomarker analysis — Correlative studies
Other: enzyme-linked immunosorbent assay — Correlative studies
  Other Names: ELISA
Other: flow cytometry — Correlative studies

SUMMARY:
RATIONALE:

Vaccines made from peptides may help the body build an effective immune response to kill tumor cells. Giving booster vaccinations may make a stronger immune response and prevent or delay the recurrence of cancer.

PURPOSE:

To evaluate the efficacy of poly-ICLC + MUCI peptide vaccine in boosting the immunologic response to MUCI in patients with triple-negative BC

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy of MUC1 peptide-poly-ICLC adjuvant vaccine in boosting systemic immunity to MUC1 in women who have completed therapy for AJCC(American Joint Committee on Cancer)stage I-III 'triple-negative' [i.e., ER(-) PR(-) HER2/neu(-)] breast cancer.

SECONDARY OBJECTIVES:

I. To evaluate the safety and toxicity of the MUC1 peptide and poly-ICLC vaccine in this cohort of patients.

OUTLINE:

Patients receive MUC-1 peptide vaccine subcutaneously (SC) and poly-ICLC vaccine SC in weeks 0, 2, and 10 in the absence of disease progression or unacceptable toxicity. Some patients may receive a booster vaccine in week 52. Patients will be followed for study-related Serious Adverse Events (SAEs) for a period of 30 days after their last vaccination. If a patient experiences a SAE while participating in this study, they will be followed until the resolution of the SAE.

ELIGIBILITY:
Inclusion Criteria:

* AJCC stage I-III infiltrating adenocarcinoma of the breast who have completed standard adjuvant or neoadjuvant therapy (surgery, radiation, biologic therapy, chemotherapy) for TNBC (ER-, PR-, HER-2/neu-)
* Patients who have completed standard therapy for triple-negative inflammatory BC are eligible
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Absolute neutrophil count >= 1,000/mm^3
* Hemoglobin >= 10.0 g/dl
* Platelet count >= 100,000/mm^3
* Total bilirubin must be within normal limits
* Transaminases (aspartate aminotransferase [AST] and/or alanine aminotransferase [ALT]) may be up to 2.5 x institutional upper limit of normal (ULN) if alkaline phosphatase is =< ULN
* Alkaline phosphatase may be up to 4 x ULN if transaminases are =< ULN
* Normal creatinine and blood urea nitrogen (BUN); if abnormal, calculated creatinine clearance must be >= 60 mg/dL
* Human immunodeficiency virus (HIV)(-), antinuclear antibody (ANA)(-), hepatitis panel (-), normal thyroid function tests; these tests will be performed at the discretion of the Investigator if warranted by history or clinical presentation
* Patients must be disease-free of prior invasive malignancies for >= 5 years, with the exception of curatively-treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* All patients must have completed surgery with sentinel and/or axillary lymph node dissection according to participating institutional guidelines
* All patients must have completed adjuvant radiation therapy according to participating institutional guidelines
* All patients must have completed either adjuvant or neoadjuvant chemotherapy according to participating institutional guidelines; the choice of chemotherapy is at the discretion of the treating physician
* Women of childbearing potential must have a negative pregnancy test and must be willing to consent to using an accepted and effective barrier form method of contraception during participation in the study and for a reasonable period thereafter
* Patients must provide written informed consent

Exclusion Criteria:

* Known metastatic BC
* Radiotherapy, chemotherapy, biologic therapy, or other investigational therapy within the preceding 4 weeks
* Previous splenectomy or radiotherapy to spleen
* Coexisting or previous malignancies except carcinoma in situ of the cervix or basal cell carcinoma of the skin
* Active or uncontrolled infection
* Psychiatric, addictive, or any disorder that compromises the ability to give informed consent to participate in or to comply with the requirements of the study
* Concurrent systemic corticosteroid treatment - must be off all steroids for at least 4 weeks prior to vaccine administration
* Any condition or behavior that in the judgment of the Investigator, would compromise the patient's ability to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-08-19; Primary Completion 2013-08-29 (Actual); Study Completion 2016-01-21 (Actual)

PRIMARY OUTCOMES:
Proportion of patients showing a positive anti-MUC1 antibody response | At week 12 (2 weeks after the 3rd injection)
  Defined as a >= 2-fold enhancement from baseline anti-MUC1 antibody immunity, or for subjects with no antibody to MUC1 at baseline, any detectable antibody immunity against MUC1. To test the hypothesis of a sufficient immunologic response, we will apply a Simon's optimum 2-stage design. The proportion of patients with an immunologic response will be calculated with a 95% confidence interval using method developed for multistage clinical trials.

SECONDARY OUTCOMES:
Safety and toxicity as assessed by NCI CTC | Weeks 0, 2, 4, 10, 12, 52, and 54 and then for 30 days after completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Baar, MD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Gorodetska I, Samusieva A, Lahuta T, Ponomarova O, Socha O, Kozeretska I. Exploring New Frontiers: Alternative Breast Cancer Treatments Through Glycocalyx Research. Breast J. 2025 May 22;2025:9952727. doi: 10.1155/tbj/9952727. eCollection 2025. PMID 40443562